CLINICAL TRIAL: NCT00303836
Title: A Phase II Study Using a Peptide Vaccine With or Without Aldesleukin Following a Lymphodepleting Chemotherapy and Reinfusion of Autologous Lymphocytes Depleted of T Regulatory Lymphocytes in Metastatic Melanoma
Brief Title: Vaccine Therapy With or Without Interleukin-2 After Chemotherapy and an Autologous White Blood Cell Infusion in Treating Patients With Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02684; P6574; NCI-06-C-0028; CDR0000459683; NCI-7547; NCI-P6574; NCT00255203 (obsolete NCT alias)
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Recurrent Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — Cyclophosphamide; fludarabine phosphate; Peripheral Blood Stem Cell Transplantation; gp100 Melanoma Antigen; MART-1 Antigen; incomplete Freund's adjuvant; montanide ISA 51; Filgrastim; Granulocyte Colony-Stimulating Factor; aldesleukin; Interleukin-2

ARMS (2):
- Arm I (Experimental): Patients undergo apheresis and in-vitro depletion of T-regulatory cells. Patients then receive a nonmyeloablative, lymphocyte-depleting preparative regimen comprising cyclophosphamide IV over 1 hour on days -8 and -7 and fludarabine IV over 15-30 minutes on days -6 to -2 followed by autologous T-regulatory-depleted lymphocytes IV over 20-30 minutes on day 0. Patients receive vaccination with gp100:209-217 (210M) and MART-1:27-35 peptides emulsified in Montanide ISA-51 subcutaneously (SC) on days 0-3, 20-23, 41-44, and 62-65. Patients also receive filgrastim (G-CSF) SC beginning on day 1 and continuing until blood counts recover.
  Interventions: Drug: cyclophosphamide; Drug: fludarabine phosphate; Biological: therapeutic autologous lymphocytes; Procedure: in vitro-treated peripheral blood stem cell transplantation; Biological: gp100 antigen; Biological: MART-1 antigen; Biological: incomplete Freund's adjuvant; Biological: filgrastim
- Arm II (Experimental): Patients receive treatment as in arm I. Patients also receive high-dose IL-2 IV over 15 minutes every 8 hours on days 0-4, beginning after the lymphocyte infusion. IL-2 treatment repeats every 3 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cyclophosphamide; Drug: fludarabine phosphate; Biological: therapeutic autologous lymphocytes; Procedure: in vitro-treated peripheral blood stem cell transplantation; Biological: gp100 antigen; Biological: MART-1 antigen; Biological: incomplete Freund's adjuvant; Biological: filgrastim; Biological: aldesleukin

INTERVENTIONS:
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Biological: therapeutic autologous lymphocytes — Given IV
  Other Names: AL; Autologous Lymphocytes; autologous T cells
Procedure: in vitro-treated peripheral blood stem cell transplantation — Undergo in vitro-treated peripheral blood stem cell transplantation
  Other Names: in vitro-treated PBPC transplantation; in vitro-treated PBSC; in vitro-treated peripheral blood progenitor cell transplantation; PBPC transplantation, in vitro-treated; peripheral blood progenitor cell transplantation, in vitro-treated
Biological: gp100 antigen — Given SC
  Other Names: gp100
Biological: MART-1 antigen — Given SC
  Other Names: Antigen LB39-AA; Antigen SK29-AA; MART-1; MART-1 Tumor Antigen
Biological: incomplete Freund's adjuvant — Given SC
  Other Names: IFA; ISA-51; Montanide ISA 51
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen
Biological: aldesleukin — Given IV
  Other Names: IL-2; Proleukin; recombinant human interleukin-2; recombinant interleukin-2
  Arms: Arm II

SUMMARY:
This randomized phase II trial is studying how well giving vaccine therapy with or without interleukin-2 after chemotherapy and an autologous white blood cell infusion works in treating patients with metastatic melanoma. Vaccines made from peptides may help the body build an effective immune response to kill tumor cells. Giving vaccine therapy with interleukin-2, chemotherapy, and an autologous white blood cell infusion may be a more effective treatment for metastatic melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the ability of gp100 and MART-1 peptide vaccines with or without a high-dose interleukin-2 (IL-2), when administered after a nonmyeloablative, lymphodepleting preparative regimen and reinfusion of autologous CD25+ T-regulatory-depleted lymphocytes, to mediate tumor regression in patients with metastatic melanoma.

SECONDARY OBJECTIVES:

I. Determine the generation of antitumor lymphocytes and the rate of repopulation of CD25+ T-regulatory cells in patients treated with this regimen.

II. Determine the toxicity of this treatment regimen.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo apheresis and in-vitro depletion of T-regulatory cells. Patients then receive a nonmyeloablative, lymphocyte-depleting preparative regimen comprising cyclophosphamide IV over 1 hour on days -8 and -7 and fludarabine IV over 15-30 minutes on days -6 to -2 followed by autologous T-regulatory-depleted lymphocytes IV over 20-30 minutes on day 0. Patients receive vaccination with gp100:209-217 (210M) and MART-1:27-35 peptides emulsified in Montanide ISA-51 subcutaneously (SC) on days 0-3, 20-23, 41-44, and 62-65. Patients also receive filgrastim (G-CSF) SC beginning on day 1 and continuing until blood counts recover.

ARM II: Patients receive treatment as in arm I. Patients also receive high-dose IL-2 IV over 15 minutes every 8 hours on days 0-4, beginning after the lymphocyte infusion. IL-2 treatment repeats every 3 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 1-3 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic melanoma

  * No tumor reactive cells available for cell transfer therapy
* Measurable disease
* Previously treated with interleukin-2 (IL-2) and meets 1 of the following criteria:

  * No response (progressive disease)
  * Recurrent disease
* HLA*0201 positive
* ECOG performance status 0 or 1
* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 8.0 g/dL
* ALT and AST < 3 times upper limit of normal
* Bilirubin ≤ 2.0 mg/dL (< 3.0 mg/dL if Gilbert's disease is present)
* Creatinine ≤ 2.0 mg/dL
* Life expectancy ≥ 3 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for up to 4 months after receiving the preparative regimen
* No active systemic infections, coagulation disorders, or other major medical illnesses of the cardiovascular, respiratory, or immune system, as evidenced by a positive stress thallium or comparable test, myocardial infarction, cardiac arrhythmias, or obstructive or restrictive pulmonary disease
* No autoimmune disease (e.g., autoimmune colitis or Crohn's disease) or primary immunodeficiency disease
* No HIV positivity
* No hepatitis B or C virus positivity
* No Epstein-Barr virus negativity
* Eligible to receive high-dose IL-2, as evidenced by the following:

  * Patients ≥ 50 years of age must have a normal cardiac stress test (e.g., stress thallium, stress MUGA, dobutamine echocardiogram, or other stress test) AND LVEF ≥ 45%
  * Patients with a history of EKG abnormalities, symptoms of cardiac ischemia, or arrhythmias must have a normal cardiac stress test AND LVEF ≥ 45%
  * Patients with a prolonged history of cigarette smoking or symptoms of respiratory dysfunction must have a normal pulmonary function test, as evidenced by FEV 1 ≥ 60% of predicted
* At least 4 weeks since prior systemic therapy
* At least 6 weeks since prior nitrosourea therapy
* No concurrent systemic steroid therapy
* Recovered immune competence after prior chemotherapy or radiotherapy
* No prior gp100:209-217 or MART-1:27-35 peptide vaccine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2005-11; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Objective clinical response (CR or PR) | Up to 2 years

SECONDARY OUTCOMES:
Presence of anti-tumor T cells | Up to 2 years
Recovery of regulatory T cells | Up to 2 years
Incidence of DLTs and SAEs graded according to CTCAE version 3.0 | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven Rosenberg, Principal Investigator — National Cancer Institute Surgery Branch
Locations (1):
- National Cancer Institute Surgery Branch, Bethesda, Maryland, United States